CLINICAL TRIAL: NCT02341352
Title: Study on Children's Dental Caries Prevention and Mechanism
Brief Title: Three Measures for the Prevention of Carious Lesions in Preschool Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Occupational Disease Prevention Hospital (Other)
Responsible Party: Principal Investigator, Xi Chen, Master, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2013-8; 81371142 (Other Grant/Funding Number: National Natural Science Foundation of China); 20120633B14 (Other Grant/Funding Number: Hangzhou Science and Technology Project)
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Probiotics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): Only behavioral education for Caregiver
- fluoride varnish (Experimental): fluoride varnish every 6 months
  Interventions: Drug: fluoride varnish
- ImmunoglobulinY (Experimental): anti-S.mutans Immunoglobulin yolk for everyday use
  Interventions: Biological: Immunoglobulin Yolk
- Probiotics (Experimental): Probiotics use for 1 months
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Drug: fluoride varnish — Sodium fluoride 50mg/ml
  Other Names: Duraphat(Colgate-palmolive company)
  Arms: fluoride varnish
Biological: Immunoglobulin Yolk — anti-Streptococcus mutans IgY
  Other Names: Aoliding oral bacteriostatic spray(Hangzhou YaSheng Biotech)
  Arms: ImmunoglobulinY
Dietary Supplement: Probiotics — 2g/day，Lactobacillus rhamnosus HN001, Bifidobacterium lactis Bi-07, Bifidobacterium lactis HN019, maltodextrin, fructose, skimmed milk powder
  Other Names: Probiotics milk power(Minsheng Pharmaceutical)
  Arms: Probiotics

SUMMARY:
Analysis different measures preventive effect on carious Lesions incidence and oral microecological system change of preschool children

DETAILED DESCRIPTION:
Different caries prevention trials including fluoride vanish, IgY-passive immunotherapy and probiotics lasting 24 months were conducted with a total of 500 children aged 24 to 54 months of age in Lin'an, Zhejiang, China. The trials were cluster- domized .After obtaining parent´s informed consent, preschool children were clinical examinated according to ICDAS-Ⅱ and microbiological tested of saliva at baseline, 1m, 6m, 12m, 18m and 24m. To find the differences of caries incidence and oral microecology change in four groups, dmfs will be assessed and saliva will be analysed in experiment.

ELIGIBILITY:
Inclusion Criteria:

* preschool children in good general health
* At least 18 deciduous teeth

Exclusion Criteria:

* With major systemic disease or on long-term medication
* Not cooperative and refuse dental treatment
* With a history of extra fluoride supplement
* Take antibiotics for nearly 8 weeks

Ages: 24 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The number of new cavitated or incipient carious lesion | 24 months after first visit
  To determine whether preschool children that only with caregiver behavior education have more new caries lesion than those taken some caries preventive measures by differences in dmfs（decay，missing，filling teeth surfaces） index after 24 months dental exams.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, Principal Investigator — Department of Conservative Dentistry and Periodontics, Affiliated Hospital of Stomatology, School of Medicine, Zhejiang University
Locations (1):
- Affiliated Hospital of Stomatology, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang J, Su L, Wang Y, Deng S. Improved High-Throughput Sequencing of the Human Oral Microbiome: From Illumina to PacBio. Can J Infect Dis Med Microbiol. 2020 Dec 11;2020:6678872. doi: 10.1155/2020/6678872. eCollection 2020. PMID 33381248
- [Derived] Wang Y, Wang S, Wu C, Chen X, Duan Z, Xu Q, Jiang W, Xu L, Wang T, Su L, Wang Y, Chen Y, Zhang J, Huang Y, Tong S, Zhou C, Deng S, Qin N. Oral Microbiome Alterations Associated with Early Childhood Caries Highlight the Importance of Carbohydrate Metabolic Activities. mSystems. 2019 Nov 5;4(6):e00450-19. doi: 10.1128/mSystems.00450-19. PMID 31690590